CLINICAL TRIAL: NCT04006431
Title: Prostate Embolization in Chronically Surveyed Patients: Effectiveness of Unilateral vs. Bilateral Embolization
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2018
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2019-07

CONDITIONS: Unilateral vs Bilateral Embolization of the Prostate Arteries
MeSH Terms: interventions — Embolization, Therapeutic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: embolization — Retrospective, observational collection with division of patients into two groups according to unilateral or bilateral embolization of the porstatic arteries.

SUMMARY:
Prostate embolization is an alternative treatment to trans urethral prostate resection in the context of benign prostatic hypertrophy. This embolization treatment is also of interest in patients with chronic anuria surveyed in relation to their prostatic hypertrophy for disundation. This survey causes discomfort and urinary tract infection. It is a population with tortuous arteries, a severe atherosclerotic overload making embolizations complex and long. Often, only unilateral embolization is possible. The purpose of this study is to compare the effectiveness in terms of disundation of unilateral vs. bilateral embolization of the prostatic arteries

DETAILED DESCRIPTION:
Prostate embolization is an alternative treatment to trans urethral prostate resection in the context of benign prostatic hypertrophy. This embolization treatment is also of interest in patients with chronic anuria surveyed in relation to their prostatic hypertrophy for disundation. This survey causes discomfort and urinary tract infection. It is a population with tortuous arteries, a severe atherosclerotic overload making embolizations complex and long. Often, only unilateral embolization is possible. The purpose of this study is to compare the effectiveness in terms of disundation of unilateral vs. bilateral embolization of the prostatic arteries.

Method of observation or investigation chosen:

Retrospective, observational collection with division of patients into two groups according to unilateral or bilateral embolization of the porstatic arteries.

Origin and nature of the data Patient's medical record: imaging stored in the PACS to confirm unilateral or bilateral embolization, perform measurements of prostate volume, urological medical record to see the effectiveness of embolization in terms of disundation, comfort of life, tolerance of embolization, effectiveness in terms of urination (IPSS score)

Data flow mode:

Data stored in redcap.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (>70 years old)
* with contraindications to surgery,
* with a chronic urinary catheterization

Exclusion Criteria:

* <70 years old
* without contraindications to surgery
* without chronic urinary catheterization

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly patients (>70 years of age) with contraindications to surgery, chronically probed
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
the effectiveness of embolization | at one month
  International prostate score symptomsScore

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Result] Frandon J, Belaouni A, Pellerin O, Thiounn N, Serrand C, Droupy S, Petitpierre F, Vernhet-Kovacsik H, Murez T, Vidal V, Ghelfi J, Pagnoux G, Codas R, de Forges H, Beregi JP, Sapoval M. Efficacy and safety of prostate artery embolization for patients with lower urinary tract symptoms and indwelling urinary catheter: A retrospective multicenter study. Diagn Interv Imaging. 2022 Dec;103(12):601-606. doi: 10.1016/j.diii.2022.07.002. Epub 2022 Aug 10. PMID 35963778